CLINICAL TRIAL: NCT03201289
Title: Microvolt T-wave Alternans in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Other Study IDs: MTWA
Record Dates: First submitted 2017-06-16; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Complications; Electrocardiogram: Electrical Alternans
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery

SUMMARY:
The purpose of this study is to measure MTWA in the patients undergoing cardiac surgery and to investigate the relation between MTWA and adverse clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients underwent cardiac surgery including coronary artery bypass graft surgery with or without cardiopulmonary bypass, cardiac valve surgery, cardiac mass excision, thoracic aorta surgery, etc.

Exclusion Criteria:

* unavailability of the recording equipment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
in hospital mortality | up to 3 months(during hospital stay)
  in hospital death

SECONDARY OUTCOMES:
postoperative complication | up to 3 months(during hospital stay)
  The secondary end points were myocardial infarction, ventricular tachycardia, atrial fibrillation, cardiogenic shock, stroke, coma, renal failure, respiratory failure, and length of stay in intensive care unit (ICU) and hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea